CLINICAL TRIAL: NCT07211776
Title: A Multicenter, Double-blinded, Randomized, Placebo Controlled Phase 3 Trial to Evaluate the Efficacy and Safety of ZL-1109 in Chinese Participants With Thyroid Eye Disease (TED)
Brief Title: A Study to Assess the Efficacy and Safety of ZL-1109 in Chinese Participants With Active Thyroid Eye Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZL-1109-002
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Eye Disease (TED)
Keywords: Thyroid Eye Disease (TED)
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of the three study arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, Investigator, Outcomes Assessor and Sponsor will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Randomized controlled period: ZL-1109 every 4 weeks (Experimental): Participants will receive ZL-1109 per protocol defined dosing regimen.
  Interventions: Drug: ZL-1109 (VRDN-003)
- Randomized controlled period: ZL-1109 every 8 weeks (Experimental): Participants will receive ZL-1109 and placebo per protocol defined dosing regimen.
  Interventions: Drug: ZL-1109 (VRDN-003); Drug: Placebo
- Randomized controlled period: Placebo every 4 weeks (Placebo Comparator): Participants will receive placebo per protocol defined dosing regimen.
  Interventions: Drug: Placebo
- OLE treatment period: ZL-1109 every 4 weeks (Other): Participants who not responded would receive ZL-1109 per protocol defined dosing regimen.
  Interventions: Drug: ZL-1109 (VRDN-003)

INTERVENTIONS:
Drug: ZL-1109 (VRDN-003) — ZL-1109 subcutaneous injection
  Arms: OLE treatment period: ZL-1109 every 4 weeks; Randomized controlled period: ZL-1109 every 4 weeks; Randomized controlled period: ZL-1109 every 8 weeks
Drug: Placebo — Matching placebo subcutaneous injection
  Arms: Randomized controlled period: Placebo every 4 weeks; Randomized controlled period: ZL-1109 every 8 weeks

SUMMARY:
A Multicenter, Double-blinded, Randomized, Placebo-controlled Phase 3 Study of ZL-1109 in Chinese Participants with Thyroid Eye Disease (TED)

DETAILED DESCRIPTION:
This is a multicenter, Phase 3, randomized, double-blinded, placebo-controlled study to evaluate the efficacy, safety and tolerability of ZL-1109 in participants with active TED. The study will comprise a screening period of up to 28 days, a double-blinded randomized placebo-controlled period of 24 weeks and an extension period. For responders and non-responders who do not want to receive open-label treatment, the study period is 52 weeks from the first dose. For non-responders who consent to and are considered eligible to receive open-label treatment, the study period is 70 weeks from the first dose.

ELIGIBILITY:
Key Inclusion Criteria:

1. Have moderate to severe TED
2. Must meet the clinical diagnosis criteria of active TED
3. Must agree to use highly effective contraception as specified in the protocol
4. Female TED participants must have a negative serum pregnancy test at screening

Key Exclusion Criteria:

1. Have received prior treatment with another anti-IGF-1R mAb or anti-thyroid stimulating hormone receptor (TSHR) mAb.
2. Have received systemic corticosteroids or steroid eye drops for any condition, or other immunosuppressive drugs for any condition, including TED, or radioactive iodine (RAI) treatment within a certain period prior to first dose.
3. Have corneal decompensation in the study eye unresponsive to medical management.
4. Have a pre-existing ophthalmic in the study eye which in the opinion of the Investigator, would confound interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-03-14 (Estimated); Study Completion 2028-01-29 (Estimated)

PRIMARY OUTCOMES:
Proptosis Responder Rate in the study eye | At Week 24
  Proportion of participants with a ≥2 mm reduction from baseline in proptosis in the study eye [without a corresponding increase of ≥2 mm in the fellow eye]

SECONDARY OUTCOMES:
Change from baseline in proptosis in the study eye | At Week 24
  Change from baseline in proptosis in the study eye
Overall Responder Rate in the study eye | At Week 24
  Proportion of participants with a ≥2 mm reduction from baseline in proptosis in the study eye [without a corresponding increase of ≥2 mm in the fellow eye]) AND ≥ 2 points reduction in CAS from baseline in the study eye [without a corresponding increase of ≥2 points in the fellow eye]
Change from baseline in Clinical Activity Score (CAS) in the study eye | At Week 24
  Change from baseline in CAS in the study eye [range, 0 to 7, with higher scores indicating greater level of inflammation]
Proportion of participants with a Clinical Activity Score (CAS) of 0 or 1 in the study eye | At Week 24
  Proportion of participants with a CAS of 0 or 1 in the study eye
Diplopia Responder Rate for participants with baseline Diplopia Score greater than 0 | At Week 24
  Proportion of participants with a reduction in Diplopia Score of ≥1 from baseline (for participants with baseline Diplopia Score greater than 0)
Diplopia Resolution Rate for participants with baseline Diplopia Score greater than 0 | At Week 24
  Proportion of participants with a reduction in Diplopia Score to 0 from baseline (for participants with baseline Diplopia Score greater than 0)
Clinical Activity Responder Rate in the study eye | At Week 24
  Clinical Activity Responder Rate in the study eye (i.e., ≥ 2 points reduction in CAS from baseline in the study eye [without a corresponding increase of ≥2 points in the fellow eye])

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - Site01006, Beijing
  - Site01009, Beijing
  - Site01010, Beijing
  - Site01029, Bengbu
  - Site01020, Changsha
  - Site01022, Chengdu
  - Site01031, Chongqing
  - Site01011, Dalian
  - Site01008, Foshan
  - Site01004, Fuzhou
  - Site01007, Guangzhou
  - Site01027, Guiyang
  - Site01018, Hangzhou
  - Site01002, Hefei
  - Site01024, Jinan
  - Site01005, Luoyang
  - Site01017, Nanchang
  - Site01001, Shanghai
  - Site01012, Shenyang
  - Site01023, Taiyuan
  - Site01013, Tianjin
  - Site01016, Wuxi
  - Site01028, Xi'an
  - Site01025, Xuzhou
  - Site01026, Yangzhou
  - Site01019, Zhengzhou
  - Site01030, Zhengzhou

IPD SHARING:
Plan to Share IPD: No
The study team does not plan to make individual participant data underlying the published results publicly available. This decision is based on two key considerations: (1) the absence of informed consent at the participant level for reuse of data beyond the pre-specified analyses outlined in the study protocol; (2) applicable privacy regulations in relevant jurisdictions which restrict the further dissemination of personally identifiable information. Aggregate-level data supporting the primary findings of the study will be made available through supplementary materials accompanying the publication, and may also be shared upon reasonable request to the corresponding author for purposes such as meta-analysis or regulatory review, provided that a formal data use agreement is executed.